CLINICAL TRIAL: NCT05677022
Title: Evaluation of the Interest of a Postural and Functional Analysis for the Follow-up of the Adapted Motor Activity of Patients Treated for Breast Cancer
Acronym: APECS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A03091-40
Record Dates: First submitted 2022-12-19; First posted 2023-01-10 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, longitudinal, single-center, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted motor activity (Experimental)
  Interventions: Other: Adapted motor activity

INTERVENTIONS:
Other: Adapted motor activity — 15-month adapted motor activity program based on a postural and functional analysis

SUMMARY:
The goal of this clinical trial is to evaluate the acceptability by patients treated for breast cancer of an adapted motor activity program over a period of 15 months controlled by a postural and functional analysis..

Participant population/health conditions: patients with newly operated breast cancer who are candidates for an adapted physical activity program

DETAILED DESCRIPTION:
This is a prospective, longitudinal, single-center, open-label study of a population of newly operated breast cancer patients who were candidates for an adapted motor activity program.

All included patients will be followed for a period of 15 months. Participating physicians will have the opportunity to recruit their patients during the 24 months following the study's initiation. The study will be completed once the last included patient has a final evaluation. The total duration of the study is 39 months (24 months of recruitment and 15 months of follow-up).

Each patient will be assessed four times: at inclusion before initiation of cancer treatment, and at M3, M9 and M15. At each patient visit with the investigating physician, an assessment will be completed on the electronic CRF by the physician or by the site CRA under the responsibility of the investigating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman, having given her consent to participate in the study,
* Patient with non-metastatic breast cancer,
* Cancer to be treated by surgery with or without adjuvant treatment (radiotherapy and/or chemotherapy).

Exclusion Criteria:

* Contraindication to the practice of a physical activity,
* Mental deficiency or any other reason that could hinder the understanding or the strict application of the protocol,
* Patient not affiliated to the French social security system,
* Patient under legal protection, guardianship or curatorship,
* Patient already included in another therapeutic study protocol aimed at evaluating the benefits of adapted physical activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of compliance | Month 15
  Patients will be considered compliant if they have attended more than 50% of the physical adaptation program sessions

SECONDARY OUTCOMES:
Assessment of the functional impact of the disease | Month 3
  The Primus is used to establish a score during the performance of a movement. The number and nature of the movements evaluated are independent from one patient to another, nevertheless 4 very precise movements will be carried out in all the patients included in this study: ironing, vacuuming, driving and the hand-grip. The tests performed on the same patient will be strictly identical from one examination to the next.
  A Primus score will be calculated for each gesture. A global score will be calculated for each patient. It corresponds to the total score obtained by the patient divided by the number of tests performed.
  For each test and for the global score, the score recorded at Day 0 will constitute the reference value. The evolution of the scores during the follow-up will be expressed as a percentage of variation in relation to this basal score.
Assessment of the functional impact of the disease | Month 9
  The Primus is used to establish a score during the performance of a movement. The number and nature of the movements evaluated are independent from one patient to another, nevertheless 4 very precise movements will be carried out in all the patients included in this study: ironing, vacuuming, driving and the hand-grip. The tests performed on the same patient will be strictly identical from one examination to the next.
  A Primus score will be calculated for each gesture. A global score will be calculated for each patient. It corresponds to the total score obtained by the patient divided by the number of tests performed.
  For each test and for the global score, the score recorded at D0 will constitute the reference value. The evolution of the scores during the follow-up will be expressed as a percentage of variation in relation to this basal score.
Assessment of the functional impact of the disease | Month 15
  The Primus is used to establish a score during the performance of a movement. The number and nature of the movements evaluated are independent from one patient to another, nevertheless 4 very precise movements will be carried out in all the patients included in this study: ironing, vacuuming, driving and the hand-grip. The tests performed on the same patient will be strictly identical from one examination to the next.
  A Primus score will be calculated for each gesture. A global score will be calculated for each patient. It corresponds to the total score obtained by the patient divided by the number of tests performed.
  For each test and for the global score, the score recorded at D0 will constitute the reference value. The evolution of the scores during the follow-up will be expressed as a percentage of variation in relation to this basal score.
Postural evaluation | Month 3
  The postural evaluation will be carried out using a force platform with strain gauges as sensors, allowing to measure the moment of the vertical force exerted on the plate, and to locate the center of pressure of the feet and to record the variations on the antero-posterior and lateral axes.
  The dual-tray platform used in the study allows separate assessment of the forces exerted under each of the lower limbs.
Postural evaluation | Month 9
  The postural evaluation will be carried out using a force platform with strain gauges as sensors, allowing to measure the moment of the vertical force exerted on the plate, and to locate the center of pressure of the feet and to record the variations on the antero-posterior and lateral axes.
  The dual-tray platform used in the study allows separate assessment of the forces exerted under each of the lower limbs.
Postural evaluation | Month 15
  The postural evaluation will be carried out using a force platform with strain gauges as sensors, allowing to measure the moment of the vertical force exerted on the plate, and to locate the center of pressure of the feet and to record the variations on the antero-posterior and lateral axes.
  The dual-tray platform used in the study allows separate assessment of the forces exerted under each of the lower limbs.
Pain assessment | Month 3
  Pain intensity will be assessed using a simple numerical scale (SNS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Pain assessment | Month 9
  Pain intensity will be assessed using a simple numerical scale (SNS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Pain assessment | Month 15
  Pain intensity will be assessed using a simple numerical scale (SNS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Functional and mobility assessment of the shoulder | Month 3
  This evaluation will be carried out using the Constant questionnaire composed of 11 questions grouped into 4 items (pain, activities of daily living, mobility and power of the shoulder). A global score ranging from 0 to 100 is obtained (almost no function to normal function).
Functional and mobility assessment of the shoulder | Month 9
  This evaluation will be carried out using the Constant questionnaire composed of 11 questions grouped into 4 items (pain, activities of daily living, mobility and power of the shoulder). A global score ranging from 0 to 100 is obtained (almost no function to normal function).
Functional and mobility assessment of the shoulder | Month 15
  This evaluation will be carried out using the Constant questionnaire composed of 11 questions grouped into 4 items (pain, activities of daily living, mobility and power of the shoulder). A global score ranging from 0 to 100 is obtained (almost no function to normal function).
Assessment of the emotional impact of the disease | Month 3
  The emotional impact of the disease will be more precisely evaluated by the HAD questionnaire, a screening tool for the most common manifestations of anxiety and depressive disorders to be completed by the patient. The scale consists of 14 questions, with 7 items assessing anxiety and 7 items assessing depression. A minimum score of 10 on one of the sub-scores was retained as a screening criterion for depressive or anxious manifestations.
Assessment of the emotional impact of the disease | Month 9
  The emotional impact of the disease will be more precisely evaluated by the HAD questionnaire, a screening tool for the most common manifestations of anxiety and depressive disorders to be completed by the patient. The scale consists of 14 questions, with 7 items assessing anxiety and 7 items assessing depression. A minimum score of 10 on one of the sub-scores was retained as a screening criterion for depressive or anxious manifestations.
Assessment of the emotional impact of the disease | Month 15
  The emotional impact of the disease will be more precisely evaluated by the HAD questionnaire, a screening tool for the most common manifestations of anxiety and depressive disorders to be completed by the patient. The scale consists of 14 questions, with 7 items assessing anxiety and 7 items assessing depression. A minimum score of 10 on one of the sub-scores was retained as a screening criterion for depressive or anxious manifestations.
Assessment of the impact of the disease on quality of life | Month 3
  Patients' quality of life will be assessed by completing the EORTC Core Quality of Life Questionnaire EORTC QLQ-C30 questionnaire with 30 questions
Assessment of the impact of the disease on quality of life | Month 3
  Patients' quality of life will be assessed by completing the EORTC Core Quality of Life Questionnaire EORTC QLQ-Br 23 module with 23 additional questions.
Assessment of the impact of the disease on quality of life | Month 9
  Patients' quality of life will be assessed by completing the EORTC Core Quality of Life Questionnaire EORTC QLQ-C30 questionnaire with 30 questions
Assessment of the impact of the disease on quality of life | Month 9
  Patients' quality of life will be assessed by completing the EORTC Core Quality of Life Questionnaire EORTC QLQ-Br 23 module with 23 additional questions.
Assessment of the impact of the disease on quality of life | Month 15
  Patients' quality of life will be assessed by completing the EORTC Core Quality of Life Questionnaire EORTC QLQ-C30 questionnaire with 30 questions.
Assessment of the impact of the disease on quality of life | Month 15
  Patients' quality of life will be assessed by completing the EORTC Core Quality of Life Questionnaire EORTC QLQ-Br 23 module with 23 additional questions.
Assessment of sarcopenia | Month 15
  Sarcopenia will be measured by impedancemetry. The parameters collected will be in kilograms.
Assessment of sarcopenia | Month 15
  Sarcopenia will be measured by impedancemetry. The parameters collected will be in percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Clairval Hospital Center, Marseille, France

IPD SHARING:
Plan to Share IPD: No